CLINICAL TRIAL: NCT06374797
Title: Auxora for the Treatment of AKI and Modulation of Injurious "Crosstalk" With the Lung: A Randomized Control Trial (KOURAGE)
Brief Title: A Study of Auxora in Patients With AKI and Injurious Lung "Crosstalk"
Acronym: KOURAGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMZ-207
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: AKI; Acute Kidney Injury; Auxora
MeSH Terms: conditions — Acute Kidney Injury | interventions — zegocractin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Auxora (Experimental)
  Interventions: Drug: Auxora
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Auxora — 1.25 mL/kg (2.0 mg/kg of zegocractin) intravenously (IV) over 4 hours at 0 hours, and then 1.0 mL/kg (1.6 mg/kg of zegocractin) IV over 4 hours at 24, 48, 72 and 96 hours for a total of 5 doses.
  Arms: Auxora
Drug: Placebo — 1.25 mL/kg IV over 4 hours at 0 hours and then 1.0 mL/kg IV over 4 hours at 24, 48, 72, and 96 hours for a total of 5 doses.
  Arms: Placebo

SUMMARY:
Approximately 150 patients with acute kidney injury (AKI) associated with acute hypoxemic respiratory failure (AHRF) will be randomized at up to 40 sites. Patients will be randomly assigned to either Auxora or matching placebo. Study drug infusions will occur every 24 hours for five consecutive days for a total of five infusions.

DETAILED DESCRIPTION:
This double blind, randomized, placebo-controlled study will evaluate the efficacy, safety, and tolerability of Auxora in patients with severe AKI who have associated AHRF. The definition of AKI and the stages of AKI will be based on the classification system proposed by the Acute Kidney Injury Working Group of Kidney Disease: Improving Global Outcomes (KDIGO) and incorporate both serum creatinine and urine volume criteria. AHRF will be defined as a P/F ≤ 300 that has been determined by either an arterial blood gas or imputed from the oxygen saturation (SpO2) recorded using pulse oximetry and is being treated with high flow nasal cannula with minimum flow rate ≥ 30 liters/min, or non-invasive mechanical ventilation, or invasive mechanical ventilation. Approximately 150 patients with severe AKI, defined as having developed either stage 2 or 3 AKI at the time of consent, who have associated AHRF will be randomized 1:1 into either the Auxora or placebo group using a computer-generated randomization scheme accessed through an interactive voice/web response system (IXRS). Randomization will be stratified by the use of invasive mechanical ventilation and by Stage 3 AKI.

Patients who are randomized to the Auxora group will receive 1.25 mL/kg (2.0 mg/kg of zegocractin) IV over 4 hours at 0 hours and then 1.0 mL/kg (1.6 mg/kg of zegocractin) IV over 4 hours at 24, 48, 72, and 96 hours for a total of 5 doses. Patients who are randomized to the placebo group will receive 1.25 mL/kg IV over 4 hours at 0 hours and then 1.0 mL/kg IV over 4 hours at 24, 48, 72, and 96 hours for a total of 5 doses. Placebo will be a matching emulsion without the active pharmaceutical ingredient zegocractin. The sponsor, investigators, pharmacists, and patients will be blinded to the assigned group. The Start of First Infusion of Study Drug (SFISD) should occur no more than 24 hours of the patient or legally authorized representative (LAR) providing informed consent. A study physician or appropriately trained delegate will perform study-specific hospital assessments immediately prior to the SFISD, and then every 24 hours after the SFISD until 720 hours (Day 30), or until discharge if earlier. All patients, including those that are discharged from the hospital to home, or to a skilled nursing facility, or to an extended care facility, will be assessed at Day 90.

All AKI should be managed according to the KDIGO 2012 guidelines which recommends maintaining adequate organ perfusion, avoiding volume overload, avoiding hyperglycemia, discontinuing nephrotoxic agents, and adjusting dosing of renally excreted medications. AHRF/acute respiratory distress syndrome (ARDS) should be managed according to the 2023 European Society of Intensive Care Medicine (ESICM) major recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 years of age.
2. The patient has developed Stage 2 or Stage 3 AKI.
3. The patient has a documented partial pressure of oxygen [Pa02]/fraction of inspired oxygen [FiO2] (P/F) ≤ 300 in the prior 24 hours, either imputed from SpO2 or obtained from an arterial blood gas, that is not explained by cardiogenic pulmonary edema or volume overload
4. The patient is being treated with either high flow nasal cannula with minimum flow rate ≥ 30 liters/min, or non-invasive mechanical ventilation, or invasive mechanical ventilation at time of randomization.
5. A female patient of childbearing potential who is sexually active with a male partner is willing to practice acceptable methods of birth control for 30 days after the last dose of study drug.
6. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 30 days after the last dose of study drug. A male patient must not donate sperm for 30 days after the last dose of study drug.
7. The patient is willing and able to, or has a legally authorized representative (LAR) who is willing and able to, provide informed consent to participate and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. The patient has a do not intubate directive.
2. The patient has chronic lung disease that requires supplemental non-invasive oxygen as an outpatient or home mechanical ventilation. The use of non-invasive mechanical ventilation to treat obstructive sleep apnea is not an exclusion.
3. The patient has been hospitalized in the ICU for more than 10 days.
4. The patient has been receiving invasive mechanical ventilation for > 120 hours.
5. The patient is receiving extracorporeal membrane oxygen (ECMO).
6. The patient has started or is planned to start kidney replacement therapy (KRT) before randomization.
7. The patient has a serum triglyceride level ≥ 500 mg/dL.
8. The patient has a direct bilirubin level >3.0 mg/dL or both a direct bilirubin level ≥ 2.0 mg/dL and an international normalized ratio (INR) ≥ 1.7.
9. AKI is suspected to be secondary to: renal artery or renal vein thrombosis; hepato-renal syndrome; cholesterol emboli syndrome; acute glomerulonephritis; vasculitis; acute allergic interstitial nephritis; intrarenal or extrarenal urinary tract obstruction; use of immune checkpoint inhibitor.
10. The patient has a known history of an organ transplant.
11. The patient has a known history of HIV infection.
12. The patient has known history of hepatitis B infection.
13. The patient is currently receiving chemotherapy.
14. The patient is currently receiving immunosuppressive medications
15. The patient is known to be pregnant or is currently nursing.
16. The patient is allergic to eggs.
17. The patient is currently participating in another study of an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Days alive, ventilator-free and kidney replacement therapy (KRT)-free from SFISD through Day 30 | SFISD through Day 30
  The primary efficacy analysis will apply the win ratio method and the Finkelstein-Schoenfeld method to the primary endpoints. The win ratio method allocates all Auxora and placebo pairs to the components that comprise the primary endpoint in a hierarchical fashion.
  Categories (a) and (c) represent Auxora wins based on all-cause mortality and days ventilator-free and KRT-free. Similarly, categories (b) and (d) represent placebo wins. Category (e) represents ties.
  (a) Death on placebo, but alive on Auxora at day 30 (b) Death on Auxora, but alive on placebo at day 30 (e) Death on placebo and death on Auxora at day 30
  If alive on placebo and alive on Auxora at day 30:
  (c) Greater number of days alive, ventilator-free and KRT-free on Auxora (d) Greater number of days alive, ventilator-free and KRT-free on Placebo (e) Equal number of days alive, ventilator-free and KRT-free We will calculate the overall win ratio by adding (a) + (c) and dividing it by the sum of (b) + (d).

SECONDARY OUTCOMES:
Major adverse kidney event (MAKE) 90-1: ≥25% decline in estimated glomerular filtration rate (eGFR) from baseline, incident KRT, and all-cause mortality at 90 days | At Day 90
MAKE 90-2: ≥35% decline in eGFR from baseline, incident KRT, and all-cause mortality at 90 days | At Day 90
Proportion of patients alive at Day 30 | At Day 30
Proportion of patients alive at Day 90 | Day 90
Days alive and ventilator-free from start of first infusion of study drug (SFISD) through Day 30 | SFISD through Day 30
Days alive and KRT-free from SFISD through Day 30 | SFISD through Day 30
Proportion of patients recovered from AHRF through Day 30 as categorized by an 8-point ordinal scale | SFISD through Day 30
  The measurement tool is an 8-point ordinal scale: 1=Death; 2=Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation(ECMO); 3=Hospitalized, requiring non-invasive ventilation or high flow supplemental oxygen; 4=Hospitalized, requiring low flow supplemental oxygen; 5=Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care; 6=Hospitalized, not requiring supplemental oxygen or ongoing medical care; 7=Discharged, requiring supplemental oxygen; 8=Discharged, not requiring supplemental oxygen
Proportion of patients receiving KRT at Day 30 | At Day 30
Proportion of patients receiving KRT at Day 90 | At Day 90
Number of patients with treatment-related adverse events (TEAE) | SFISD through Day 90
Number of patients with grade 3 TEAEs | SFISD through Day 90

OTHER OUTCOMES:
Days alive and not hospitalized through Day 30 | SFISD through Day 30
Proportion of patients re-hospitalized through Day 30 | SFISD through Day 30
Proportion of patients re-hospitalized through Day 90 | SFISD through Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Chief Medical Officer, Study Director — CalciMedica, Inc.
Locations (34):
- United States (34):
  - University of Alabama, Birmingham, Alabama
  - Chandler Regional Hospital, Chandler, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA, Los Angeles, California
  - Stanford Health Care, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Tampa General, Tampa, Florida
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - St Luke's Hospital, Boise, Idaho
  - Northwestern University-Pulmonary & Critical Care Medicine, Chicago, Illinois
  - University of Indiana, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Brigham & Woman's Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford, Detroit, Michigan
  - My Michigan Health, Midland, Michigan
  - University of Missouri, Columbia, Missouri
  - Hannibal Regional, Hannibal, Missouri
  - Holy Name, Teaneck, New Jersey
  - NYU Langone Health - Brooklyn, Brooklyn, New York
  - NYU Langone Health - Bellview, New York, New York
  - NYU Langone Health - Tisch Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - UT Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia